CLINICAL TRIAL: NCT05982483
Title: Erector Spinae Plane Block vs. Usual Care for ED Patients With Mechanical Back Pain: A Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block vs. Usual Care for ED Patients With Mechanical Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Island Health (Other)
Responsible Party: Principal Investigator, Ben Ho, Emergency department staff physician, Island Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C2018-102
Record Dates: First submitted 2023-07-06; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Back Pain
Keywords: nerve block; back pain; regional anaesthesia; analgesia
MeSH Terms: conditions — Back Pain; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants in both cohorts had pink chlorhexidine skin prep and a dressing applied to the back. Research team members performing the telephone follow-up were blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP cohort (Experimental): Randomized to receive the ultrasound-guided ESP block.
  Interventions: Procedure: Erector Spinae plane block using 20 ml of bupivicaine 0.25%
- Usual care cohort (Active Comparator): Randomized to usual care as dictated by the treating emergency physician
  Interventions: Drug: Usual care

INTERVENTIONS:
Procedure: Erector Spinae plane block using 20 ml of bupivicaine 0.25% — Utilizing the in line approach, a 22 gauge 3.5" spinal needle was guided the the tip of the transverse process corresponding to the area of maximal tenderness or central to the reported area of spasm. 1% lidocaine with epinephrine was used for skin anaesthesia and for hydro-localization of the needle tip on approach to the tip of the transverse process. Once the needle tip made contact with the transverse process, 2-3 ml of 1% lidocaine with epinephrine was injected to open the ESP plane. If there was no reported tachycardia after approximately 45 seconds, 20 ml of 0.25% bupivicaine was injected into the ESP plane.
  Arms: ESP cohort
Drug: Usual care — Analgesia as dictated by the treating emergency physician
  Arms: Usual care cohort

SUMMARY:
The goal of this clinical trial is to compare the Erector Spinae plane (ESP) block, a nerve block, to usual care in emergency department patients with back pain. The main question it aims to answer:

Is the ESP block superior to usual care in the treatment of back pain in the emergency department? Participants will be randomly assigned to the ESP or the usual care group. Pain improvement at the time of emergency department discharge will be compared.

ELIGIBILITY:
Inclusion Criteria: Patients deemed to have mechanical back pain with a component of paravertebral tenderness or paravertebral spasm reported by the patient or noted on examination by treating physician.

Exclusion Criteria:

* previous recipient of erector spinae plane block
* exam concerning for cauda equina syndrome
* current IV drug use
* organ transplant recipient
* history of or suspected bleeding diathesis
* current use of anticoagulants
* sepsis or soft tissue infection at site of the block within last three months
* pregnancy
* overt malignancy involving skin or underlying soft tissue at the site of block
* allergy to any of the research medications
* inability to participate in telephone follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Numeric Verbal Pain Score (NVPS) reduction at emergency department discharge | Numeric verbal pain score (NVPS) at time of randomization compared with NVPS at time of discharge from the emergency department up to 24 hours after randomization.
  The NVPS is an 11-point verbal pain scale from 0 to 10 with 0 representing no pain and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
Number of patients requiring post randomization Emergency department (ED) opiate analgesia analgesia use | Time of randomization to time of ED discharge up to 24 hours after randomization.
  Opiate medication dose and route of administration was recorded
Emergency department (ED) length of stay. | Time of ED triage to time of ED discharge up to 24 hours after triage.
  Time spent in the emergency department.
Brief Pain Inventory (BPI) score reduction from baseline | Time of randomization compared to 1 day, 1 week, 1 month, and 3 months post Emergency department visit
  The Brief Pain Inventory (BPI) is widely used to measure a patients' pain intensity and interference the pain has on daily function measured in 7 categories: mood, work, general activity, walking, relationships, enjoyment of life, and sleep. The patient rates each of these on a scale from 0-10with 0 representing no interference and 10 complete interference in that aspect of life. The initial BPI was recorded at time of randomization and subsequent BPI's recorded by telephone follow-up at predetermined time intervals
Number of patients requiring post Emergency department discharge opiate analgesia use | Date of randomization to 1 day after randomization, 1 day after randomization to 1 week after randomization, 1week after randomization to 1 month after randomization, 1 month after randomization to 3 months after randomization.
  During telephone follow up, patients were asked if there was any opiate analgesia used during the pre-determined time period.
Post Emergency department (ED) discharge Numeric Verbal Pain Score (NVPS) | 1 day after randomization, 1 week after randomization, 1 month after randomization, 3 months after randomization.
  At telephone follow up at predetermined time intervals, patients were asked what their most severe level of pain they were currently experiencing as measured by the NVPS
Number of patients able to ambulate post ED treatment if unable to on ED admission | Time of ED triage compared to time of ED discharge up to 24 hours after triage.
  If patient was unable to ambulate on ED admission, did ED treatment allow ambulation without assistance: yes or no
Number of patients requiring Emergency department (ED) return visits for back pain | Date of randomization to 1 day after randomization, 1 day after randomization to 1 week after randomization, 1week after randomization to 1 month after randomization, 1 month after randomization to 3 months after randomization.
  At telephone follow up at predetermined intervals, patients were asked if they had to return subsequently to the emergency department due to their back pain

CONTACTS AND LOCATIONS:
Locations (1):
- Nanaimo Regional General Hospital, Nanaimo, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho B, Fyfe-Brown R, Chopra S, McMeel K. The erector spinae plane block vs. usual care for treatment of mechanical back pain in the emergency department: a pilot study. CJEM. 2024 Aug;26(8):543-548. doi: 10.1007/s43678-024-00748-7. Epub 2024 Jul 31. PMID 39083200